CLINICAL TRIAL: NCT01426542
Title: Pilot Study of Topiramate Prophylaxis in Infants Undergoing Surgery for Congenital Heart Disease
Brief Title: Preventing Brain Injury in Infants With Congenital Heart Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 216534
Record Dates: First submitted 2011-08-05; First posted 2011-08-31 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Cyanotic Congenital Heart Disease
Keywords: brain injury; stroke; cerebral palsy; seizures
MeSH Terms: conditions — Brain Injuries; Stroke; Cerebral Palsy; Seizures | interventions — Topiramate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topiramate (Experimental)
  Interventions: Drug: Topiramate
- Control (Active Comparator): These infants will undergo surgery, but will not receive topiramate
  Interventions: Other: No medication, but routine heart surgery

INTERVENTIONS:
Drug: Topiramate — Topiramate 5 mg/kg by mouth (or by feeding tube) once a day for one week before and one week after heart surgery.
  Arms: Topiramate
Other: No medication, but routine heart surgery — No medication, but routine heart surgery
  Arms: Control

SUMMARY:
Newborn babies with congenital heart disease often require surgery in the first month of life. The risks of brain damage from congenital heart disease and from the various corrective surgeries are high because of poor levels of oxygen reaching the brain. Topiramate is an anti-convulsant medication that protects brain cells from damage due to low amounts of oxygen in animal studies. The investigators hypothesize that giving topiramate to babies with congenital heart disease before and after surgery will decrease the amount of brain damage caused by the heart disease and/or the surgery to correct the heart disease.

DETAILED DESCRIPTION:
Infants with cyanotic congenital heart disease undergoing surgery in the neonatal period have a high rate of brain injury resulting in seizures, stroke, cerebral palsy, and neurodevelopmental delays. Neuroimaging abnormalities are found in 30% to 60% of cases and neurodevelopmental impairments occur in more than half of these children. The mechanisms of brain injury in these children are not fully understood. Experimental animal models have shown that the abundant release of glutamate in the brain during hypoxic-ischemic insult results in brain injury. Blocking glutamate receptors by administration of the anticonvulsant topiramate has been shown to prevent such injury in animal studies. This study is an open pilot trial of peri-operative topiramate administration to infants with cyanotic congenital heart disease to test the feasibility of this approach and generate preliminary data about markers of brain injury (serum S100B levels and urine metabolomics) and neurodevelopment at 18 months of age. If the approach is feasible and the preliminary data are encouraging a larger efficacy trial will be designed. Although topiramate has been used in neonates and infants to treat seizures and in a pilot study in term infants with hypoxic-ischemic encephalopathy, this is the first study of its effects on markers of brain injury and neurologic outcomes in infants with cyanotic congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 2 months
* Cyanotic congenital heart disease requiring surgery

Exclusion Criteria:

* Genetic syndromes with high risk of neurodevelopmental delay
* Gestational age less than 35 weeks at birth
* Multiple organ failure or multiple organ anomalies

Max Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Plasma S100B | 1 week before surgery, 1 day and 1 week after surgery
  Baseline plasma S100B levels will be determined prior to surgery (at enrollment) with repeat levels at the two timepoints after surgery. Main outcome will be change from baseline.

SECONDARY OUTCOMES:
Mullen Scales of Early Learning | 18 months of age
  This broad assessment of neurodevelopment includes five scales: Gross Motor, Visual Reception, Fine Motor, Expressive Language, and Receptive Language, with further testing if needed to explore deficits.
Changes from baseline in urine metabolomics | 1 week before surgery, 1 day and 1 week after surgery
  Urine specimens obtained at enrollment and at the two time points after surgery will be assessed for a broad range of metabolites (complex molecules). Changes from baseline will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Underwood, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Children's Hospital, Sacramento, California, United States